CLINICAL TRIAL: NCT06190301
Title: Safety and Efficacy of Intralesional Rituximab Injection Versus Involved Site Radiation Therapy in Primary Ocular Adnexal MALT Lymphoma: a Multicenter Randomized Controlled Trial
Brief Title: RCT on Intralesional Rituximab Injection Versus ISRT in Ocular Adnexal MALT Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong Lu, Professor, MD, PhD, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023KYPJ125-3
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Primary Ocular Adnexal MALT Lymphoma
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralesional Rituximab Injection (Experimental)
  Interventions: Drug: Rituximab
- Involved Site Radiation Therapy (Active Comparator)
  Interventions: Radiation: Involved Site Radiation Therapy

INTERVENTIONS:
Drug: Rituximab — Intralesional Rituximab Injection
  Arms: Intralesional Rituximab Injection
Radiation: Involved Site Radiation Therapy — Involved Site Radiation Therapy
  Arms: Involved Site Radiation Therapy

SUMMARY:
This project proposes to establish a prospective, multicenter, randomized, controlled clinical study to compare the safety and efficacy of Intralesional Rituximab Injection versus Involved Site Radiation Therapy for the treatment of primary ocular adnexal MALT lymphoma. The aim is to provide high-level clinical evidence for the treatment of ocular adnexal MALT lymphoma and to offer patients treatment options that have fewer complications and comparable therapeutic effects.

ELIGIBILITY:
Inclusion criteria

1. Age between 18 to 75 years old.
2. Ocular adnexal MALT lymphoma with a comprehensive diagnosis based on pathology, clinical manifestations, and biological characteristics according to the WHO classification of tumors of hematopoietic and lymphoid tissues.
3. Based on the TNM staging of ocular adnexal lymphoma, patients with stages T1-3 of ocular adnexal MALT lymphoma without involvement of intraconal compartment are included.
4. Willing to participate the trial and sign the informed consent form.

Exclusion criteria

1. Based on the TNM staging of ocular adnexal lymphoma (Table 1), patients staged as T2/T3 with involvement of intraconal compartment and patients staged as T4.
2. Patients who have previously received local or systemic radiation, chemotherapy, or drug treatment specifically for ocular adnexal MALT lymphoma.
3. Presence of cataract and is anticipated to require surgical treatment within a certain period after enrollment; existing cataract affects visual field testing and fundoscopic examination; vision affected by cataract is <20/40.
4. In addition to the need for treatment of ocular adnexal MALT lymphoma, there is a requirement for other ocular procedures (e.g., full-thickness corneal transplant or retinal surgery) or an anticipated need for another emergent ocular surgery.
5. Complicated with other ocular diseases: including corneal abnormalities or existing corneal infections, iridocorneal endothelial syndrome, anterior segment dysgenesis, true microphthalmos, uveitis, glaucoma, ocular trauma, and retinal disorders such as central retinal vein occlusion, central retinal artery occlusion, retinal detachment, etc.
6. The statue of HBV or HIV infection.
7. Need for long-term use of local or systemic steroids.
8. Patients already enrolled in other drug clinical trials.
9. Pregnant or breastfeeding women.
10. Serious systemic diseases: advanced cardiac disease, kidney disease, respiratory disease, or other malignant tumors, etc.
11. Inability to understand the research content.

If both eyes of a patient meet the inclusion criteria, the right eye will be selected for participation in the study, while the left eye will receive the same treatment, but its data will not be included in this research. Each patient can have only one eye participating in the study. If both eyes of a patient meet the inclusion criteria and the patient is randomized to the ISRT group, the eye with the larger lesion or with more symptomatic disease is treated first, and in the case of well tolerability, the other eye is irradiated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The cumulative occurrence rate of complications of grade ≥2 within 5 years after treatment commencement | within 5 years after treatment commencement

SECONDARY OUTCOMES:
overall response rate | within 5 years after treatment commencement
progression-free survival | within 5 years after treatment commencement
time to next treatment | within 5 years after treatment commencement
overall survival | within 5 years after treatment commencement

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Access Criteria: Available upon reasonable request

REFERENCES:
- [Derived] Liu Y, Gao Y, Jin L, Li Q, Wang X, Wu Y, Zhou J, Liu W, Wang L, Dong Y, Zheng Y, Chen L, Li J, Su S, Tang J, Wang Y, Huang W, Cheng C, Li C, An N, Tan J, Chen H, Guo H, Wang Y, Zhou Q, Han F, Liu H, Zhu Y, Lu R. Safety and efficacy of intralesional rituximab injection versus involved site radiation therapy in primary ocular adnexal MALT lymphoma: study protocol for a multicentre randomised controlled trial. BMJ Open. 2024 Nov 27;14(11):e084904. doi: 10.1136/bmjopen-2024-084904. PMID 39608989